CLINICAL TRIAL: NCT04527952
Title: The Fasting and Shifted Timing (FAST) of Eating Study
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Brie Turner-McGrievy, Associate Professor, University of South Carolina
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00089911
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Overweight and Obesity
Keywords: fasting
MeSH Terms: conditions — Overweight; Obesity; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Time-restricted feeding (TRF) (Experimental): Participants will eat the majority of their calories in the day. More specifically participants will consume 70% of their total calories before 5 pm and the remaining 30% after 5 pm.
  Interventions: Behavioral: Online handouts describing how to follow each diet for 1 week each
- Intermittent fasting (IF) (Active Comparator): This involves eating all of one's meals within a specific time (e.g. 8 hours) frame and fasting for the remaining hours (16 hours) in a day.
  Interventions: Behavioral: Online handouts describing how to follow each diet for 1 week each
- Alternate day fasting (ADF) (Active Comparator): This involves complete fasting (i.e. no food or caloric containing beverages, only water consumption) for roughly an entire 36-hour period, followed by an ad libitum feeding day.
  Interventions: Behavioral: Online handouts describing how to follow each diet for 1 week each

INTERVENTIONS:
Behavioral: Online handouts describing how to follow each diet for 1 week each — Participants will receive handouts via email about how to follow each diet

SUMMARY:
The aim of this study is to assess peoples' satisfaction with their diet based on adhering to three different meal-timing protocols for one week each: (1) Time-restricted feeding (TRF); (2) Intermittent fasting (IF); and (3) Alternate day fasting (ADF). The overall goal of this study is to determine if people would find it easy or difficult to follow these diet protocols for the purpose of weight management.

DETAILED DESCRIPTION:
Fasting and time-restricted feeding (TRF) have become increasingly popular in nutrition research due to the potential health benefits they may provide. Several animal studies, and more recently some human studies, have indicated regular meal-timing (i.e. eating mostly in the day) or fasting have been beneficial for controlling weight, blood pressure, cholesterol, glucose, and insulin sensitivity.

These types of eating patterns may offer the same "anti-aging" health benefits as traditional caloric restriction (i.e. consistent and routine adherence to a very low-calorie diet).While caloric restriction is considered the gold standard for weight management, weight regain often limits the long-term effectiveness of this approach. People often experience increases in hunger, which make it difficult to sustain this type of behavior.Therefore, researchers are turning to these dietary approaches as alternatives to low-calorie diets in an effort to obtain the same benefits, but with less burden on participants.

However, it is not clear if the adherence to these types of diet protocols are any better than a low-calorie diet. Would people be more satisfied with meal-timing or fasting over a traditional very low-calorie diet? That is the main research question of this study.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Have a BMI between 25 - 49.9 kg/m2.
* Have a scale at home, or some way of weighing yourself regularly, so that you can report your body weight to the research staff.
* Be able to check emails regularly, because all of the surveys need to be completed online.

Exclusion Criteria:

* NOT be already practicing any of these fasting approaches.
* NOT currently diagnosed with diabetes.
* NOT taking any appetite suppressants or prescription weight loss medications.
* NOT planning on getting pregnant within the next 6 weeks.
* Do NOT currently have any eating disorders.
* Have NOT lost or gained a significant amount of weight (i.e. 10 pounds or more) within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Weight loss-week 1 | 1 week
  We will assess weight loss via self-report after 1 week on diet #1
Weight loss- week 2 | 1 week
  We will assess weight loss via self-report after 1 week on diet #2
Weight loss- week 3 | 1 week
  We will assess weight loss via self-report after 1 week on diet #3

SECONDARY OUTCOMES:
Energy intake-week 1 | 6 weeks
  Energy (kcal) intake will be assessed after 1 week on diet #1
Energy intake- week 2 | 6 weeks
  Energy (kcal) intake will be assessed after 1 week on diet #2
Energy intake- week 3 | 6 weeks
  Energy (kcal) intake will be assessed after 1 week on diet #3

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle Turner-McGrievy, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner-McGrievy GM, Wirth MD, Bernhart JA, Aydin H. The Fasting and Shifted Timing (FAST) of Eating Study: A pilot feasibility randomized crossover intervention assessing the acceptability of three different fasting diet approaches. Appetite. 2022 Sep 1;176:106135. doi: 10.1016/j.appet.2022.106135. Epub 2022 Jun 16. PMID 35716852